CLINICAL TRIAL: NCT00141843
Title: A Randomized Two-Way Blinded Crossover-Design Study to Establish the Bioequivalence of B-Domain Deleted Recombinant Factor VIII (BDDrFVIII,Refacto AF) With a Full Length Recombinant Factor VIII Preparation (FLrFVIII,Advate), Followed by an Open-Label Trial of the Safety and Efficacy of ReFacto AF in Previously Treated Patients With Hemophilia A.
Brief Title: Study to Establish Bioequivalence of ReFacto AF (BDDrFVIII) With Advate (FLrFVIII) in Hemophilia A
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Wyeth is now a wholly owned subsidiary of Pfizer (Industry)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Prevention
Other Study IDs: 3082B2-310
Record Dates: First submitted 2005-08-30; First posted 2005-09-01 (Estimated); Last update posted 2008-04-22 (Estimated); Status verified 2008-04

CONDITIONS: Hemophilia A
Keywords: Hemophilia A
MeSH Terms: conditions — Hemophilia A | interventions — Factor VIII; recombinant factor VIII SQ

INTERVENTIONS:
Genetic: ReFacto AF
Genetic: B-Domain deleted Recombinant Factor VIII
Genetic: BDDrFVIII

SUMMARY:
The study will consist of two parts: a safety and efficacy period in which all subjects will participate and a pharmacokinetic analysis period, in which 30 eligible subjects will participate to compare ReFacto AF and Advate bioequivalency and safety and efficacy of ReFacto AF in patients with Hemophilia A.

ELIGIBILITY:
Inclusion Criteria:

* Male subjects with severe or moderately severe hemophilia A
* A negative past medical history of a Factor VIII inhibitor
* Age greater than or equal to 12 years

Exclusion Criteria:

* A history of Factor VIII inhibitors
* Presence of a bleeding disorder in addition to hemophilia
* Known hypersensitivity to hamster protein

Min Age: 12 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 100
Dates: Start 2005-07; Primary Completion 2006-11 (Actual); Study Completion 2006-11 (Actual)

PRIMARY OUTCOMES:
To determine the incidence rate of Factor VIII inhibitors in the study patient population.To establish bioequivalence of ReFacto AF as compared to Advate using the one stage Factor VIII activity assay.

SECONDARY OUTCOMES:
To characterize the efficacy of ReFActo AF in preventing and treating bleeding episodes during prophylaxis.To characterize PK of ReFacto AF as compared to Advate over time.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Wyeth is now a wholly owned subsidiary of Pfizer; Trial Manager, Principal Investigator — For Germany, MedInfoDEU@wyeth.com; Trial Manager, Principal Investigator — For Italy, descresg@wyeth.com; Trial Manager, Principal Investigator — For Australia, New Zealand, medinfo@wyeth.com; Trial Manager, Principal Investigator — For Netherlands, trials-NL@wyeth.com; Trial Manager, Principal Investigator — For Sweden, Finland,MedInfoNord@wyeth.com; Trial Manager, Principal Investigator — For Hungary, WPBUMED@wyeth.com; Trial Manager, Principal Investigator — For Poland, WVWZMED@wyeth.com; Trial Manager, Principal Investigator — For Belgium, trials-BEL@wyeth.com
Locations (41):
- United States (21):
  - Phoenix, Arizona
  - Sacramento, California
  - San Diego, California
  - Aurora, Colorado
  - Atlanta, Georgia
  - Iowa City, Iowa
  - New Orleans, Louisiana
  - Worcester, Massachusetts
  - East Lansing, Michigan
  - St Louis, Missouri
  - New Brunswick, New Jersey
  - Buffalo, New York
  - New Hyde Park, New York
  - Chapel Hill, North Carolina
  - Dayton, Ohio
  - Hershey, Pennsylvania
  - Philadelphia, Pennsylvania
  - Nashville, Tennessee
  - Houston, Texas
  - Salt Lake City, Utah
  - Charlottesville, Virginia
- Perth, Australia
- Leuven, Belgium
- Helsinki, Finland
- France (2):
  - Le Kremlin-Bicêtre
  - Rouen
- Germany (2):
  - Berlin
  - Münster
- Budapest, Hungary
- Milan, Italy
- Groningen, Netherlands
- New Zealand (2):
  - Auckland
  - Hamilton
- Poland (4):
  - Lodz
  - Poznan
  - Warsaw
  - Wroclaw
- Spain (2):
  - Madrid
  - Valencia
- Sweden (2):
  - Malmo
  - Stockholm